CLINICAL TRIAL: NCT02238548
Title: Effect of Raw Milk on the Immune Response Upon Cholera Vaccination
Acronym: MOSAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL49042.081.14
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Infection
Keywords: immunity; vaccination; milk
MeSH Terms: conditions — Infections | interventions — Dukoral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Placebo Comparator): Regular cholera vaccination
  Interventions: Biological: Cholera vaccination
- Milk bolus (Experimental): Cholera vaccination - raw milk - bolus
  Interventions: Biological: Cholera vaccination; Other: Raw milk
- Milk controlled (Experimental): Cholera vaccination - raw milk - controlled intake
  Interventions: Biological: Cholera vaccination; Other: Raw milk

INTERVENTIONS:
Biological: Cholera vaccination — Oral cholera vaccination on day 0 and day 14
  Other Names: Dukoral
Other: Raw milk
  Arms: Milk bolus; Milk controlled

SUMMARY:
Rationale: Infections are an important worldwide cause of death, both in elderly and young children. Therefore, support of immunity could help to reduce the incidence of infections. To screen the potential of specific foods or food ingredients to support immunity, oral vaccination can serve as a model. In this study, oral cholera vaccination will be applied in human adult volunteers, and used as a model to study the support of the immune response by raw milk.

Objective: To investigate whether raw milk is able to enhance the immune response as induced by oral cholera vaccination.

Study design: The study is designed as a single-blind randomized controlled trial of 4 weeks.

Study population: Healthy subjects of 18-50 years of age.

Intervention: Raw milk, obtained from farms that comply to the high quality requirements for production of raw milk, and that has been screened according to the safety criteria for raw milk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 yr
* Signed informed consent
* Availability of internet connection
* Male or female
* Willing to stop blood donation at the blood bank during the study period

Exclusion Criteria:

* Currently participating in another clinical trial
* Previous Cholera, Salmonella, or E. coli vaccination
* Tonsillectomy
* Acute gastroenteritis in the past 2 months
* Use of antibiotics in the past 2 months
* Hypersensitivity to the vaccine, to formaldehyde or to any of the excipients (sodium salts)
* Pregnancy or lactating (pregnancy test will be performed on the vaccination days)
* Not willing to drink raw milk
* Allergic to milk or lactose-intolerant
* Disease of GI tract, liver, gall bladder, kidneys, thyroid gland
* Immune-compromised
* Use of immunosuppressive drugs
* Drug abuse, and not willing/able to stop this during the study
* Excessive alcohol usage (men: >4 consumptions/day or >20 consumptions/week; women: >3 consumptions/day or >15 consumptions/week)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in cholera toxin-specific IgA and IgG antibody level in nasal wash as a marker of the vaccination response | baseline and day 18

SECONDARY OUTCOMES:
Change in the cholera toxin-specific IgA and IgG antibody level in serum as a marker of the vaccination response | baseline and day 18
Change in the cholera toxin-specific IgA antibody level in feces as a marker of the vaccination response | baseline and day 28
Change in the cholera toxin-specific IgA and IgG antibody level in saliva as a marker of the vaccination response | baseline and day 18
Change in the expression of tissue homing markers on IgA and IgG antibody-secreting B cells in peripheral blood as markers of the route of modulation of the vaccination response | baseline and day 18
Cholera toxin-specific T cell proliferation as marker of modulation of the vaccination response | baseline and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Els van Hoffen, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Netherlands